CLINICAL TRIAL: NCT02201082
Title: Evaluation of the Timing of the Nebulization Related to the Physiotherapy Session
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Physionebu
Record Dates: First submitted 2014-02-20; First posted 2014-07-25 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nebulization and airway clearance technique (Experimental): nebulization combined to airway clearance
  Interventions: Procedure: Airway clearance technique; Drug: Amikacin nebulization
- Nebulization (Active Comparator): nebulization
  Interventions: Drug: Amikacin nebulization

INTERVENTIONS:
Procedure: Airway clearance technique
  Arms: Nebulization and airway clearance technique
Drug: Amikacin nebulization

SUMMARY:
The purpose of this study is to determine the optimal time for the nebulization depending on the respiratory physiotherapy session in cystic fibrosis patients.

ELIGIBILITY:
Inclusion Criteria:

* Stable cystic fibrosis patients older than 16 y.o.
* Pseudomonas aeruginosa colonization
* Hypersecretion

Exclusion Criteria:

* Kidney failure
* No pregnancy

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2012-09; Primary Completion 2013-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Urinary excretion of amikacin | 24h after the nebulization
  Pharmacokinetic study of the urinary excretion of amikacin after nebulization

SECONDARY OUTCOMES:
Amikacin concentration into the sputum | At the end of the nebulization, an expected average of 20 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium